CLINICAL TRIAL: NCT03260244
Title: A Clinical Evaluation Using EnSite Precision Cardiac Mapping System (Software Version 2.0.1 or Higher) in a Real-World Environment
Brief Title: EnSite Precision Observational Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10159
Record Dates: First submitted 2017-07-05; First posted 2017-08-24 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Arrhythmia
Keywords: atrial fibrillation; atrial flutter; supraventricular tachycardia; ventricular tachycardia; premature ventricular contractions; cardiac mapping system
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter; Tachycardia, Supraventricular; Tachycardia, Ventricular; Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Procedure: cardiac mapping and radiofrequency ablation procedure — It is a minimally invasive procedure which can be performed using either general or conscious sedation. During catheter ablation, catheters (narrow, flexible tubes) are inserted into a blood vessel, often through a site in the groin (upper thigh) or neck, and guided through the vein until they reach the heart. Small electrodes on the tip of the catheters stimulate and record the heart's activity. This test, called an electrophysiology study (EPS), allows the doctor to pinpoint the exact location of the short circuit. Another word for pinpointing the exact location of the short circuit is 'mapping', for which precision is a key requirement to maximize a successful outcome.
  Once the location is confirmed, the short circuit is either destroyed (to reopen the electrical pathway) or blocked (to prevent it from sending faulty signals to the rest of the heart).

SUMMARY:
This document is a clinical investigation plan (CIP) for the EnSite Precision Observational Study.

This clinical study is intended to quantify and characterize the usage of the EnSite Precision™ Cardiac Mapping System (Software version 2.0.1 or higher) in a real-world environment. This study will be conducted in patients who are indicated for a cardiac electrophysiological (EP) mapping and radio frequency ablation procedure using a three-dimensional system.

DETAILED DESCRIPTION:
The EnSite Precision™ Cardiac Mapping System is a newly developed system that introduces features such as Delayed Enhancement Magnetic Resonance Imaging (DE-MRI) image integration, lesion marking automaticity, automatic mapping, and workflow flexibility to aid in the success of complex ablation procedures. Utilization of this system in the treatment of complex ablation procedures and its impact on patient outcomes is not well characterized. This clinical study is designed to collect a broad range of usage scenarios, therefore this clinical study has limited patient selection criteria and data collection is focused on EnSite Precision™ Cardiac Mapping System usage and patient outcomes.

The data collected from the procedure (performed per Instructions For Use (IFU) and per standard practice of the physician) as well as the 12 month follow up period enables the Sponsor to review the system's standard practice usage. This information will be added to the current knowledge and understanding of treatment options for patients with arrhythmias, which can assist the Sponsor to provide future recommendations for best practices to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for a cardiac electrophysiology mapping and radiofrequency ablation procedure using a 3-dimensional mapping system per Instructions for Use
* Over 18 years of age
* Able to provide informed consent for study participation and willing and able to comply with the protocol described evaluations and follow up schedule

Exclusion Criteria:

* Patients who are only presenting with:

  * Atrioventricular Nodal Reentrant Tachycardia (AVNRT)
  * Atrioventricular Reentrant Tachycardia (AVRT)
* Planned cryoablation procedure
* Implanted with a neurostimulator
* Contraindication to anticoagulation
* Known presence of cardiac thrombus
* Recent (<3 months) myocardial infarction or unstable angina or coronary artery by-pass
* Currently enrolled in a clinical study/investigation evaluating another device or drug that would confound the results of this study
* Pregnant or nursing
* Individuals whose willingness to volunteer in a study, in the judgement of investigator or public authorities, could be unduly influenced by lack of or loss of the autonomy due to immaturity, or mental disability, or adverse personal circumstances, or hierarchical influence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended population for this clinical study is patients over the age of 18 years who are eligible for a cardiac electrophysiology mapping and radiofrequency ablation procedure using the EnSite Precision™ Cardiac Mapping System.
Sampling Method: Probability Sample
Enrollment: 1065 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, PhD, Study Director — Abbott
Locations (7):
- United States (7):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Cardiology Associates of North East Arkansas, Jonesboro, Arkansas
  - Arkansas Cardiology, Little Rock, Arkansas
  - Bethesda Memorial Hospital, Boynton Beach, Florida
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Aurora Medical Group, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: All subjects enrolled in the study.
Period: Overall Study
Arm/Group | All Subjects
Started | 1065
Treated | 925
1-month Follow up | 898
6-month Follow up | 765
12-month Follow up | 722
Completed | 779
Not Completed | 286
Not completed — Death | 19
Not completed — Lost to Follow-up | 60
Not completed — Withdrawal by Subject | 48
Not completed — Procedure Not Performed | 21
Not completed — Enrollment Criteria Not Met | 31
Not completed — Procedure Not Performed Per Protocol | 12
Not completed — Subject Noncompliance | 6
Not completed — No inducible Arrhythmia | 2
Not completed — Procedure Not Performed by Trained Physician on Study | 2
Not completed — Screen Failure | 2
Not completed — Treated Off Label | 69
Not completed — No Radiofrequency Ablation | 14

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 925
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 279
  Male | 646
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 751
  Canada | 174

OUTCOME MEASURES:

1. Primary Outcome: Rate of Acute Success Based on Pre-defined Procedural Endpoints
Description: The number and proportion of subjects with acute success will be summarized. Acute success was defined as the physician's goal or intention for the procedure.
Time Frame: during procedure
Population: Analysis Population, number of subjects ablated per study protocol
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 925
Participants | 901

2. Primary Outcome: Freedom From Arrhythmia Recurrence
Description: This analysis will be performed using the Kaplan-Meier (KM) analyses. The start date is the date of the index procedure. For subjects who do not experience an event, their follow up duration will be defined from the start date to the date of death, withdrawal, or last follow-up, whichever occurred later.
Time Frame: From date of procedure until the date of first documented arrhythmia recurrence or date of study completion or withdrawal for any cause, whichever came first, assessed up to 12 months
Population: Subjects who completed the 12-month visit post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 722
Participants | 471

ADVERSE EVENTS:
Time Frame: No adverse event data were collected during the procedure. No adverse event data were collected during the 12 month follow-up.
Description: Adverse Events were not collected during this clinical study.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 20/1065
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data and results from the clinical investigation are the sole property of the Sponsor. The Investigators will not use this clinical investigation-related data without the written consent of the Sponsor for any purpose other than for clinical investigation completion or for generation of publication materials, as referenced in the Clinical Trial Agreement. Single-center results are not allowed to be published or presented before the multi-center results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03260244/Prot_SAP_000.pdf